CLINICAL TRIAL: NCT01457365
Title: Vitamin D Status and Its Correlation to Bone Density, Bone Turnover Markers and Muscle Function in Community-dwelling People in Sichuan Province , P.R. China
Brief Title: Vitamin D Deficiency Epidemiological Research in Sichuan, China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Decai Chen, Professor, West China Hospital
Other Study IDs: IISP-VDCHINA
Record Dates: First submitted 2011-10-17; First posted 2011-10-21 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- subjects: it is a cross-sectional research and there is only one group.

SUMMARY:
Vitamin D insufficiency and deficiency is pandemic in the world.Sichuan Basin has a subtropical monsoon climate with China's lowest sunshine totals. Inferably, the prevalence of vitamin D insufficiency/deficiency in Sichuan basin is high, and possibly the highest in China. This study will research the serum 25OHD level to get the prevalence of vitamin D deficiency and insufficiency of urban and rural residents in Sichuan Province, China.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 30 years old living in Sichuan province.

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In total, 1500 female subjects aged more than 30 years old (750 urban and 750 rural females) will be included
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-02 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Serum 25OHD | 0 day.
  It is a cross-sectional study. All measurements will be performed once after subjects are enrolled.
serum calcium and phosphate, creatinine, PTH, BALP and CTX | 0 day
  It is a cross-sectional study. All measurements will be performed once after subjects are enrolled.
Bone mineral density of lumbar spine and hip | 0 day.
  It is a cross-sectional study. All measurements will be performed once after subjects are enrolled.
Short physical performance battery | 0 day.
  It is a cross-sectional study. All measurements will be performed once after subjects are enrolled.

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital, Sicuhuan University, Chengdu, Sichuan, China